CLINICAL TRIAL: NCT06114407
Title: Baricitinib in the Treatment of Refractory Axial Spondyloarthritis Patients: A Comparison With Tofacitinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Healthcare Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Samaresh Das, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4548
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Spondyloarthritis, Axial
Keywords: Spondyloarthritis; Tofacitinib; Baricitinib; Refractory; Axial
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylarthritis | interventions — baricitinib; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Participants of 'Baricitinib' arm will be treated with tablet baricitinib 2 mg twice daily for 12 weeks
  Interventions: Drug: Baricitinib 2mg
- Tofacitinib (Active Comparator): Participants of 'Tofacininib' arm getting tablet tofacitinib 5 mg twice daily for 12 weeks will be taken as historical control arm from another study on the efficacy of tofacitinib in refractory axial spondyloarthritis
  Interventions: Drug: Tofacitinib 5 mg

INTERVENTIONS:
Drug: Baricitinib 2mg — Participants of arm 'A' will be treated with tablet baricitinib 2 mg twice daily for 12 weeks
  Other Names: Baritinib 2 mg
  Arms: Baricitinib
Drug: Tofacitinib 5 mg — Participants of arm 'B' getting tablet tofacitinib 5 mg twice daily for 12 weeks will be taken as historical control arm from another study on the efficacy of tofacitinib in refractory axial spondyloarthritis
  Other Names: Tofacent 5 mg
  Arms: Tofacitinib

SUMMARY:
Axial Spondylarthritis (ax-SpA) is an important cause of inflammatory back pain in young adults. Janus kinase inhibitors (JAKi) has been approved for treatment of ax-SpA. Tofacitinib and baricitinib are drugs from same family (JAKi). Baricitinib is relatively less expensive than Tofacitinib.

The goal of this non-inferiority clinical trial is to learn about the efficacy of baricitinib in refractory axial spondyloarthritis ( ax-SpA) and to compare its effect with that of tofacitinib. The main questions it aims to answer are:

1. Is baricitinib 4 mg effective in refractory ax-SpA?
2. Is baricitinib non-inferior to tofacitinib in refractory ax-SpA? Participants (treatment group, 92 patients) will be treated with baricitinib 2 mg twice daily for 12 weeks. Ninety two patients getting tofacitinib 10 mg/day (comparison group) will be taken as historical control from another study on the efficacy of tofacitinib in refractory ax-SpA?

DETAILED DESCRIPTION:
This clinical trial will be conducted in the department of Rheumatology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka from October 2023-March 2025. A total of 184 patients of both genders (age ≥18 years) with refractory ax-SpA meeting the inclusion and exclusion criteria will be enrolled in this study after having informed written consent. There will be two groups with 92 patients in each group. Treatment group (92 patients) will get baricitinib 4 mg daily. Ninety two patients getting tofacitinib 10 mg/day (control arm) will be taken as historical control from another ongoing study in this department. Patients of refractory ax-SpA with high disease activity (ASDAS-CRP≥2.1) will be the entry criteria in this study.

At baseline CBC, ESR, CRP, SGPT, Serum creatinine and X-ray SI joint (A/P view), HLA-B27(if needed), CXR P/A view and MT test, fasting lipid profile will be done. Baricitinib will be given to patients free of cost. Drug adherence will be ensured by monthly pill count. Follow up visit will be done at 4th and 12th week. At each follow up patients will be evaluated clinically, relevant laboratory test and will be assessed for any side effects. All the findings will be noted in a semi-structure questionnaire. At 12th week patients will be evaluated for efficacy. Outcome will be assessed by ASDAS CRP and a change of ≥ 1.1 units from baseline for clinically important improvement and≥ 2.0 units for major improvement. Disease activity will also be assessed by ASDAS-ESR, BASDAI, functional assessment by BASFI, spinal mobility by BASMI, pain, stiffness and patient global assessment by NRS, enthesitis byMASES, quality of life by Bangla version of SF-36, Bangla version of HAQ-DI and pilot Bangla version of ASQoL. Chi-square test will used for analysis of categorical variables. Comparison of the two groups will be done using independent t-test when the data are in normal distribution and Man-Whitney U test in case of skewed distribution. At 95% confidence interval P value < 0.05 will be considered statistically significant.

Each patient will be informed about the nature and purpose of the study. This study will be free from any undue benefits or influences. If any serious adverse events develop, drugs will be stopped and the patients will be treated with utmost care. Privacy, anonymity and confidentiality of every patient will be maintained in every step. Every patient will have the rights to participate and withdraw from the study at any point of time. The withdrawal of the patients will not alter their deserved medical care. Ethical clearance will be taken from Institutional Review Board (IRB) of BSMMU.

If baricitinib is found effective in refractory ax-SpA, it will decrease the treatment cost of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients meeting the ASAS classification criteria for axial spondyloarthritis
3. Patients fulfilling the definition of refractory axial spondyloarthritis
4. Patients with ASDAS-CRP ≥ 2.1

Exclusion Criteria:

1. Patients who are currently on treatment or had been previously treated with bDMARDs or tsDMARDS (including JAK inhibitors)
2. Hemoglobin < 9 gm/dl
3. WBC count < 4000/cmm, Neutrophil count < 1000 cmm, Platelet count < 100000/cmm
4. Any current or previous history of serious opportunistic infection including tuberculosis
5. Live vaccine within 3 months prior to the first dose
6. GFR < 50 ml/min
7. ALT > 2 times upper limit normal
8. Pregnancy, breastfeeding or women of reproductive age group not using effective contraceptive
9. Current or previous history of malignancy, lymphoproliferative disease
10. New York Heart Association Class III and IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score-C Reative Protein ( ASDAS-CRP) | ASDAS CRP will be assessed at baseline, 4th and 12th week
  To calculate ASDAS-CRP, besides the value of CRP, the four other items are back pain duration of morning stiffness, peripheral pain/swelling and patient global assessment of disease activity (these are assessed by 0-10cm, visual analogue scale [VAS] or 0-10, numerical rating scale [NRS]).
  Four disease activity states were categorized by ASAS: "inactive disease", "moderate disease activity", "high disease activity" and "very high disease activity".The 3 cut-offs chosen to separate these states are: <1.3 "inactive disease", 1.3 to <2.1 "low disease activity", 2.1 to <3.5 "high disease activity" and >3.5 "very high disease activity".
  Patients of refractory ax-SpA with high disease activity (ASDAS-CRP≥2.1) will be the entry criteria in this study.
  Primary outcome will be assessed by ASDAS CRP and a change of ≥ 1.1 units from baseline for clinically important improvement and ≥ 2.0 units for major improvement.

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score-ESR ( ASDAS-ESR) | ASDAS ESR will be assessed at baseline, 4th and 12th week
  To calculate ASDAS-ESR, besides the value of ESR (mm/hr), the four other items are back pain duration of morning stiffness, peripheral pain/swelling and patient global assessment of disease activity (these are assessed by 0-10cm, visual analogue scale [VAS] or 0-10, numerical rating scale [NRS]).
  Four disease activity states were categorized by ASAS: "inactive disease", "moderate disease activity", "high disease activity" and "very high disease activity".The 3 cut-offs chosen to separate these states are: <1.3 "inactive disease", 1.3 to <2.1 "low disease activity", 2.1 to <3.5 "high disease activity" and >3.5 "very high disease activity".
  Outcome will be assessed by ASDAS ESR and a change of ≥ 1.1 units from baseline for clinically important improvement and ≥ 2.0 units for major improvement.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | BASDAI will be assessed at baseline, 4th and 12th week
  The BASDAI consists of a 01 through 10 scale (01 being no problem and 10 being worst problem) which is used to answer 6 questions pertaining to 5 major symptoms of AS: Fatigue, spinal pain, joint pain/ swelling, areas of localized tenderness ( also called enthesitis or inflammation of tendons or ligaments), morning stiffness duration, morning stiffness severity. The index results a final 0-10 BASDAI score.
Bath Ankylosing Spondylitis Functional Index (BASFI) | BASFI will be assessed at baseline, 4th and 12th week
  BASFI scores 10 items
  1. Putting on your socks or tights without help or aids (eg, sock aid).
  2. Bending forward from the waist to pick up a pen from the floor without an aid.
  3. Reaching up to a high shelf without help or aids (eg, helping hand).
  4. Getting up out of an armless dining room chair without using your hands or any other help.
  5. Getting up off the floor without help from lying on your back.
  6. Standing unsupported for 10 min without discomfort.
  7. Climbing 12 to 15 steps without using a handrail or walking aid. One foot at each step.
  8. Looking over your shoulder without turning your body.
  9. Doing physically demanding activities (eg, physiotherapy, exercises, gardening or sports).
  10. Doing a full day's activities, whether it be at home or at work. The BASFI is the mean of 10 item scores completed on a numerical rating scale. A Bangla validated version of BASFI will used in this study.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | BASMI will be assessed at baseline, 4th and 12th week
  BASMI includes five clinical measurements that reflect axial mobility:
  1. tragus to wall
  2. lumbar flexion
  3. cervical rotation
  4. lumbar side flexion
  5. intermalleolar distance.
  Grading 0-10 or linear function. Total score 0-10.
Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | MASES will be assessed at baseline, 4th and 12th week
  MASES includes enthesitis at 13 Sites:
  * Costochondral 1 right/left
  * Costochondral 7 right/left
  * Spina iliaca anterior superior right/left
  * Crista iliaca right/left
  * Spina iliaca posterior right/left
  * Processus spinosus L5
  * Achilles tendon, proximal insertion right/left. No grading All sites are scored as 0 or 1 The MASES is the sum of all site scores (from 0 to 13).
Ankylosing Spondylitis Quality of Life Questionnaire(ASQoL) | ASQoL will be assessed at baseline, 4th and 12th week
  ASQoL includes 18 questions with response 'Yes' or 'No' scoring 01 or 0 respectively.
  1. My condition limits the places I can go
  2. I sometimes feel like crying
  3. I have difficulty dressing
  4. I struggle to do jobs around the house
  5. It's impossible to sleep
  6. I am unable to join in activities with my friends/family
  7. I am tired all the time
  8. I have to keep stopping what I am doing to rest
  9. I have unbearable pain
  10. It takes a long time to get going in the morning
  11. I am unable to do jobs around the house
  12. I get tired easily
  13. I often get frustrated
  14. The pain is always there
  15. I feel I miss out on a lot
  16. I find it difficult to wash my hair
  17. My condition gets me down
  18. I worry about letting people down All item scores are added to give a total score. Scores can range from 0 (good QoL) to 18 (poor QoL).
  A Bangla version of ASQoL will be used in this study.

OTHER OUTCOMES:
Health Assessment questionnaire Disability Index (HAQ-DI) | HAQ-DI will be assessed at baseline, 4th and 12th week
  HAQ-DI includes 8 categories with 20 questions about physical abilities
  1. Dressing and Grooming
  2. Arising
  3. Eating
  4. Walking
  5. Hygiene
  6. Reach
  7. Grip
  8. Activities Each category includes aids or devices or help from another person. The higher score in each category is counted. Sum of the scores are divided by 8. A Bangla validated version of HAQ-DI will be used in this study.
36-Item Short Form Survey ( SF-36) | SF-36 will be assessed at baseline, 4th and 12th week
  SF-36 measures health related quality of life covering 8 domains of health including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Samaresh Das, M B B S, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

REFERENCES:
- [Background] Abdal SJ, Yesmin S, Shazzad MN, Azad MAK, Shahin MA, Choudhury MR, Islam MN, Haq SA. Development of a Bangla version of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and the Bath Ankylosing Spondylitis Functional Index (BASFI). Int J Rheum Dis. 2021 Jan;24(1):74-80. doi: 10.1111/1756-185X.14008. Epub 2020 Nov 1. PMID 33135389
- [Background] Baraliakos X, Kiltz U, Peters S, Appel H, Dybowski F, Igelmann M, Kalthoff L, Krause D, Menne HJ, Saracbasi-Zender E, Schmitz-Bortz E, Vigneswaran M, Braun J. Efficiency of treatment with non-steroidal anti-inflammatory drugs according to current recommendations in patients with radiographic and non-radiographic axial spondyloarthritis. Rheumatology (Oxford). 2017 Jan;56(1):95-102. doi: 10.1093/rheumatology/kew367. Epub 2016 Oct 25. PMID 27997346
- [Background] Deodhar A, Sliwinska-Stanczyk P, Xu H, Baraliakos X, Gensler LS, Fleishaker D, Wang L, Wu J, Menon S, Wang C, Dina O, Fallon L, Kanik KS, van der Heijde D. Tofacitinib for the treatment of ankylosing spondylitis: a phase III, randomised, double-blind, placebo-controlled study. Ann Rheum Dis. 2021 Aug;80(8):1004-1013. doi: 10.1136/annrheumdis-2020-219601. Epub 2021 Apr 27. PMID 33906853
- [Background] Leung YY, Lee W, Lui NL, Rouse M, McKenna SP, Thumboo J. Adaptation of Chinese and English versions of the Ankylosing Spondylitis quality of life (ASQoL) scale for use in Singapore. BMC Musculoskelet Disord. 2017 Aug 17;18(1):353. doi: 10.1186/s12891-017-1715-x. PMID 28818056
- [Background] Machado P, Landewe R, Lie E, Kvien TK, Braun J, Baker D, van der Heijde D; Assessment of SpondyloArthritis international Society. Ankylosing Spondylitis Disease Activity Score (ASDAS): defining cut-off values for disease activity states and improvement scores. Ann Rheum Dis. 2011 Jan;70(1):47-53. doi: 10.1136/ard.2010.138594. Epub 2010 Nov 10. PMID 21068095
- [Background] Machado P, Navarro-Compan V, Landewe R, van Gaalen FA, Roux C, van der Heijde D. Calculating the ankylosing spondylitis disease activity score if the conventional c-reactive protein level is below the limit of detection or if high-sensitivity c-reactive protein is used: an analysis in the DESIR cohort. Arthritis Rheumatol. 2015 Feb;67(2):408-13. doi: 10.1002/art.38921. PMID 25332195
- [Background] Miceli-Richard C, Dougados M. Tracking JAKs in spondyloarthritis: rationale and expectations. Ann Rheum Dis. 2017 Aug;76(8):1325-1326. doi: 10.1136/annrheumdis-2016-210886. Epub 2017 Mar 17. No abstract available. PMID 28314752
- [Background] Ramiro S, Nikiphorou E, Sepriano A, Ortolan A, Webers C, Baraliakos X, Landewe RBM, Van den Bosch FE, Boteva B, Bremander A, Carron P, Ciurea A, van Gaalen FA, Geher P, Gensler L, Hermann J, de Hooge M, Husakova M, Kiltz U, Lopez-Medina C, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Nissen MJ, Pimentel-Santos FM, Poddubnyy D, Proft F, Rudwaleit M, Telkman M, Zhao SS, Ziade N, van der Heijde D. ASAS-EULAR recommendations for the management of axial spondyloarthritis: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):19-34. doi: 10.1136/ard-2022-223296. Epub 2022 Oct 21. PMID 36270658
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, Dougados M, Hermann KG, Landewe R, Maksymowych W, van der Heijde D. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009 Jun;68 Suppl 2:ii1-44. doi: 10.1136/ard.2008.104018. PMID 19433414
- [Background] Smith JA, Colbert RA. Review: The interleukin-23/interleukin-17 axis in spondyloarthritis pathogenesis: Th17 and beyond. Arthritis Rheumatol. 2014 Feb;66(2):231-41. doi: 10.1002/art.38291. No abstract available. PMID 24504793
- [Background] Toussirot E. The Use of Janus Kinase Inhibitors in Axial Spondyloarthritis: Current Insights. Pharmaceuticals (Basel). 2022 Feb 22;15(3):270. doi: 10.3390/ph15030270. PMID 35337068
- [Background] Veale DJ, McGonagle D, McInnes IB, Krueger JG, Ritchlin CT, Elewaut D, Kanik KS, Hendrikx T, Berstein G, Hodge J, Telliez JB. The rationale for Janus kinase inhibitors for the treatment of spondyloarthritis. Rheumatology (Oxford). 2019 Feb 1;58(2):197-205. doi: 10.1093/rheumatology/key070. PMID 29618084
- [Background] Zahid-Al-Quadir A, Zaman MM, Ahmed S, Bhuiyan MR, Rahman MM, Patwary I, Das BB, Hossain SA, Paul S, Shahin A, Rahman M, Haq SA. Prevalence of musculoskeletal conditions and related disabilities in Bangladeshi adults: a cross-sectional national survey. BMC Rheumatol. 2020 Dec 16;4(1):69. doi: 10.1186/s41927-020-00169-w. PMID 33323124